CLINICAL TRIAL: NCT03460457
Title: Phase I Study of Tolerance and Pharmacokinetics of TQB2450 Injection
Brief Title: Tolerance and Pharmacokinetics of TQB2450
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-I-01
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 (Experimental)
  Interventions: Drug: TQB2450

INTERVENTIONS:
Drug: TQB2450 — Pharmacokinetics/Dynamics Study

SUMMARY:
To study the pharmacokinetic characteristics of TQB2450 in the human body, recommend a reasonable regimen for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignancy diagnosed with pathology or cytology who have failed standard treatment or no standard treatment;
* 18-70 years old;Eastern Cooperative Oncology Group performance status:0-1,Life expectancy of more than 3 months;
* Main organs function is normal;
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped;
* Patients should be voluntary and sign the informed consents before taking part in the study;

Exclusion Criteria:

* Patients who have received programmed cell death protein 1(PD-1) or programmed cell death protein ligand(PD-L1) antibody treatment;
* Patients who had any> 3 degree immune-related adverse event during any previous immunotherapy received;
* Appeared severe hypersensitivity after taking other monoclonal antibody drugs;
* Other malignancies have been diagnosed in the past 2 years except cured or locally curable cancers, such as cutaneous or squamous cell carcinoma, superficial bladder cancer, cervical cancer or orthotopic carcinoma of the breast;
* Known spinal cord compression, cancer meningitis patients, new onset of central nervous system metastasis or stable control of symptoms in patients with brain metastases less than 4 weeks; asymptomatic and stable imaging without the need for corticosteroid treatment；
* Patients with hypothyroidism over 2 degrees;
* Patients with active, or who have had, and are likely to relapse, autoimmune diseases; the following patients are enrolled: skin disorders without systemic treatment (eg vitiligo, psoriasis, hair loss);
* Patients treated with glucocorticoids or other immunosuppressive agents within 4 weeks prior to dosing;
* Interstitial lung disease or non-contagious pneumonia (including past history and current illness); uncontrolled systemic diseases including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc. except for radiotherapy-induced interstitial pneumonitis;
* Serious chronic or active infections require systemic antibacterial, antifungal or antiviral treatment (allowing antiviral treatment in patients with hepatocellular carcinoma), including tuberculosis infection;
* Unstable pleural effusion, pericardial effusion or ascites;
* Significant cardiovascular diseases such as heart failure of New York Heart Academy(NYHA) Class 2 and above, myocardial infarction within the past 3 months, unstable arrhythmias (including QT interval ≥480 ms) or unstable Angina;
* Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history;
* Hypertension (systolic BP ≥140 mmHg, diastolic BP ≥90 mmHg) still uncontrollable by one medication;
* Hepatitis B virus patients with active replication (DNA> 500 cps / mL), hepatitis C;
* The first medication interval from the patient: the last chemotherapy for at least 4 weeks, biological products at least five half-lives;
* The first medication interval from the patient: the last chemotherapy for at least 4 weeks, biological products at least five half-lives;
* Inoculated with vaccine or attenuated vaccine within 4 weeks before first administration;
* Major surgery, or unhealed wounds, ulcers or fractures within 4 weeks prior to the first dose;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose(MTD) | 21 days
dose-limiting toxicity(DLT) | 21 days

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax) | 21 days
Peak time（Tmax） | 21 days
Half life（t1/2） | 21 days
Area under the plasma concentration versus time curve (AUC) | 21 days
Clearance（CL） | 21 days
objective response rate(ORR) | evaluated in the end of each 3 cycles up to intolerance the toxicity or progression disease (up to 24 months)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xue J, Xue L, Tang W, Ge X, Zhao W, Li Q, Peng W, Dai C, Guo Y, Li J. TQB2450 in patients with advanced malignant tumors: results from a phase I dose-escalation and expansion study. Ther Adv Med Oncol. 2024 Jan 6;16:17588359231220516. doi: 10.1177/17588359231220516. eCollection 2024. PMID 38188467